CLINICAL TRIAL: NCT04037332
Title: Monitoring of Molecular Markers of Artemisinin Resistance in Plasmodium Falciparum Malaria: Repeated Cross-sectional Assessments in DR Congo, Nigeria and Uganda
Brief Title: Monitoring of Molecular Markers of Artemisinin Resistance Through Repeated Cross-sectional Assessments in DR Congo, Nigeria and Uganda
Acronym: Caramal DRM
Status: Completed | Type: Observational
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: Clinton Health Access Initiative, Nigeria (Other); Akena Associates Ltd. (Unknown); Kinshasa School of Public Health (Other); Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: P 001-18-2.0
Record Dates: First submitted 2019-07-25; First posted 2019-07-30 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2019-07

CONDITIONS: Severe Malaria
MeSH Terms: conditions — Malaria | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bloodspot from finger prick (performed for malaria RDT), dried on filter paper and analyzed for mutations of P. falciparum gene encoding kelch (K13)-propeller domains
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Pre-RAS roll-out . Group I: I. Children presenting directly to a referral health facility without prior administration of RAS (pre-RAS): provides a baseline assessment of artemisinin resistance marker prevalence before the introduction of RAS
  Interventions: Other: Blood sample (combined with malaria RDT) followed by gentoyping analysis
- Post-RAS roll-out - Group II: II. Children presenting directly to a referral health facility without prior administration of RAS (post-RAS): group not receiving pre-referral RAS and hence having baseline pressure for K13 resistance markers.
  Interventions: Other: Blood sample (combined with malaria RDT) followed by gentoyping analysis
- Post-RAS roll-out - Group III: III. Children receiving pre-referral RAS from community-based provider and successfully referred to a referral health facility: group receiving pre-referral RAS (monotherapy).
  Interventions: Other: Blood sample (combined with malaria RDT) followed by gentoyping analysis
- Post-RAS roll-out - Group IV: IV. Children receiving pre-referral RAS from community-based provider but not completing referral to a referral health facility, followed-up at their home on day 28: children malaria-positive on Day 28 may have an increased chance of harboring a resistant infection.
  Interventions: Other: Blood sample (combined with malaria RDT) followed by gentoyping analysis

INTERVENTIONS:
Other: Blood sample (combined with malaria RDT) followed by gentoyping analysis — Finger-prick blood samples collected from children with signs of severe febrile illness and a positive mRDT presenting to community-based providers and referral facilities ; analysis for mutations in portions of a P. falciparum gene encoding kelch (K13)-propeller domain

SUMMARY:
Currently, 16 African countries include the use of pre-referral rectal artesunate (RAS) in their treatment policies. However, guidelines for RAS use vary widely across countries and inappropriate use of RAS as a monotherapy and consequential development of resistances against artemisinin based treatments is of particular concern.

In the frame of the Unitaid-funded "Community Access to Rectal Artesunate for Malaria" (CARAMAL) Project, quality-assured RAS will be rolled in selected areas of the Democratic Republic of the Congo (DRC), Nigeria and Uganda. Approximately 3,000 treatments of RAS will be dispensed by trained community health workers to children <5 years of age in each project country per year.

Linked to the tracking of (severe) malaria patients in the frame of the CARAMAL project, this study will assess the frequency of artemisinin resistance markers in the study settings and tentatively assess whether the introduction of RAS could increase the selection of resistant P. falciparum strains. The study will be conducted in close collaboration with the Global Malaria Programme of the WHO. Finger-prick blood samples will be collected from children < 5 years of age with signs of severe febrile illness and a positive mRDT presenting to community-based providers and referral facilities before and after the pilot roll-out of pre-referral RAS at community level.

DETAILED DESCRIPTION:
Currently, 16 African countries include the use of pre-referral rectal artesunate (RAS) in their treatment policies and a number of countries have begun to implement RAS. However, guidelines for RAS use vary widely across countries and often do not align with WHO recommendations. Of particular concern in this context is the inappropriate use of RAS as a monotherapy (i.e. without subsequent ACT treatment).

In the frame of the Unitaid-funded "Community Access to Rectal Artesunate for Malaria" (CARAMAL) Project, quality-assured (QA) RAS will be rolled out through integrated Community Case Management (iCCM) schemes in selected areas of the Democratic Republic of the Congo (DRC), Nigeria and Uganda. The goal of the CARAMAL Project is to contribute to reducing malaria mortality in children by improving the community management of suspected severe malaria cases. The project will contribute to this goal by advancing the development of operational guidance to catalyse effective and appropriate scale-up of quality-assured rectal artesunate (RAS) as pre-referral treatment of severe malaria.

In the frame of the CARAMAL project, approximately 3,000 treatments of RAS will be dispensed by trained community health workers to children <5 years of age in each project country per year. Children treated with pre-referral RAS will be referred to a higher-level health facility for comprehensive clinical management, including the administration of a full course of an artemisinin-based combination therapy, as per WHO guidelines.

While phenotypic resistance of the Plasmodium parasites against artemisinin has not yet been document in the study settings, this potential threat is a major concern. The administration of artemisinin monotherapies increases drug pressure, which may lead to the selection of drug resistance conferring mutations. Mutations in portions of a P. falciparum gene encoding kelch (K13)-propeller domains are the currently known major determinant of partial resistance against artemisinin. Data on artemisinin resistance of Plasmodium parasites in the CARAMAL Project countries are patchy. K13-propeller polymorphisms previously reported from Cambodia have been found e.g. in parasites from northern Uganda, but the mutations linked to artemisinin resistance were uncommon and did not seem to increase over time. The general notion is that numerous K13 polymorphisms circulate in Africa but their distribution does not currently support the spread of artemisinin resistance.

Linked to the tracking of (severe) malaria patients in the frame of the CARAMAL project, this study will assess the frequency of artemisinin resistance markers in the study settings and tentatively assess whether the introduction of RAS could increase the selection of resistant P. falciparum strains. The study will be conducted in close collaboration with the Global Malaria Programme of the WHO. Finger-prick blood samples will be collected from children < 5 years of age with signs of severe febrile illness and a positive mRDT presenting to community-based providers and referral facilities before and after the pilot roll-out of pre-referral RAS at community level.

Dried blood spots on filter papers will be sent to a WHO-chosen laboratory (Malaria Molecular Epidemiology Unit at the Pasteur Institute in Cambodia) for molecular analyses to assess the presence of markers of artemisinin resistance (K13-propeller sequence polymorphisms).

ELIGIBILITY:
Inclusion Criteria:

* age below 5 years
* enrolled in CARAMAL Project
* history of fever plus danger signs indicative of severe febrile illness / suspected severe malaria, according to local iCCM guidelines
* positive malaria test result by RDT or microscopy
* written informed consent from a parent or guardian

Exclusion Criteria:

* no current malaria infection
* mixed or mono-infection with a non-P. falciparum species known prior to sample collection
* no permanent residence in project area

Max Age: 5 Years | Sex: All
Age Groups: Child
Study Population: All children <5 years in the Health Districts / Health Zones included into the "Community Access to Rectal Artesunate for Malaria" (CARAMAL) Project in the Democratic Republic of the Congo (DRC), Nigeria and Uganda and matching the eligibility criteria will be included
Sampling Method: Non-Probability Sample
Enrollment: 916 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
K13-propeller sequence polymorphisms in P. falciparum | Through study completion, up to one year
  Prevalence of molecular markers of artemisinin resistance in P. falciparum, namely K13-propeller sequence polymorphisms - before, after introduction of RAS in respective study area

CONTACTS AND LOCATIONS:
Overall Officials: Christian Burri, Principal Investigator — Swiss TPH, Department of Medicine; Christian Lengeler, PhD, Principal Investigator — Swiss TPH, Department of Epidemiology and Public Health
Locations (7):
- Democratic Republic of the Congo (3):
  - Health Zone of Kenge, Kenge, Kwango
  - Health Zone of Ipamu, Ipamu, Kwilu
  - Health Zone of Kingandu, Kingandu, Kwilu
- Adamawa State, selected LGAs, Yola, Adamawa, Nigeria
- Uganda (3):
  - Apac District, Lira, Apac
  - Kole District, Lira, Kole
  - Oyam District, Lira, Oyam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Registration info on major study into which drug resistance monitoring is nested — https://clinicaltrials.gov/ct2/show/NCT03568344?term=caramal&rank=1